CLINICAL TRIAL: NCT02464553
Title: EuroPainClinics® Study I (Prospective Randomized Double Blinded Trial)
Brief Title: EuroPainClinics® Study I (Prospective Trial)
Acronym: EPCSI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Patients received unplanned additional therapy during follow-up
Sponsor: Europainclinics z.ú. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 74/EK/15
Record Dates: First submitted 2015-05-26; First posted 2015-06-08 (Estimated); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: Lumbar Spinal Stenosis
Keywords: Low Back Pain Pain; Periradicular therapy; Spinal Stenosis with neurologic changes
MeSH Terms: conditions — Spinal Stenosis; Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): 1x periradicular therapy in one intervertebral space, corresponding with pain radiating dermatome
  Interventions: Other: periradicular therapy (PRT)
- Group B (Experimental): 2x periradicular therapy in two intervertebral spaces, the first corresponding with pain radiating dermatome the second according magnetic resonance visualization where stenosis is situated
  Interventions: Other: periradicular therapy (PRT)

INTERVENTIONS:
Other: periradicular therapy (PRT) — RTG controlled periradicular therapy (PRT) is a microinvasive interventional pain release procedure. Advantage of targeted pain therapy is exact administration of effective drugs to the nerve root in the area of the thoracic, lumbar or sacral spines.

SUMMARY:
In this prospective multi-centre double-blind trial the effect of the X-ray examinations controlled periradicular therapy should be examined in (approximately 300) adult patients with low back pain pain caused by foraminal stenosis radiculopathy or spinal stenosis.

A periradicular therapy (PRT) is a special radiological, low-risk therapy for chronic back pain caused by wear and tear of the cervical, thoracic, and lumbar spine or a herniated disc or disc bulge. Partially pain might also radiate to the hips or extremities and cause radicular symptoms.

DETAILED DESCRIPTION:
Controlled periradicular therapy (PRT) is a microinvasive interventional pain release procedure. Advantage of targeted pain therapy is exact administration of effective drugs to the nerve root in the area of the thoracic, lumbar or sacral spines. It is used like as effective treatment in the patients with radicular pain caused by foraminal stenosis radiculopathy or spinal stenosis.

Spinal stenosis is the narrowing of spaces in the spine which causes pressure on the spinal cord and nerves. Discogenic radicular irritation syndrome is usually caused by protrusion of intervertebral disc or prolapsed disc. The most common is lumbar and sacral radiculopathy which could by exactly verified by CT or magnetic resonance imaging. The biggest profit with the best response on this therapy has patients who are resistant for physiotherapy or per oral medicament therapy.

Intervertebral space verification is provided by X-ray examination imaging. Than in this place is Tuohy needle inserted. Position of Tuohy needle is verified by application of low dose of contrast. When the right position of needle is secured than effective drugs are administered: local anesthetic - Bupivacaine 0,25% (1-2ml) together with corticosteroid injection -Depo-Medrol (40mg). PRT involves several medicable effects: anaesthetic - positive effect on pain transmission in nerve fibers, antichemical - limitation of chemical products from sequestered discs, Anti-edematous - reduction of root nerve oedema, antiphlogistic - inhibition of phospholipase A2, antifibrotic - reduction of scar production.

Trial will compare groups of patients after fulfilment inclusion criteria's who will undergo microinvasive interventional pain release procedure - PRT.

The first group of patients will undergo PRT procedure in the intervertebral space responsible for skin dermatome were the pain is radiating.

Second group of patients will undergo double PRT procedure in the intervertebral space responsible for skin dermatome where the pain is radiating and also in the intervertebral space above where usually is disc lesion responsible for origin of pain localized. After first visit in ambulance patients will be about study informed. After agreement patient will be in to the study involved. Specific unique nine digits number will be assigned to each patient. Then patients will be randomized in to groups by special evaluated software created especially for this study. Patients will agree that about type of PRT (one level or two levels) will be informed until the end of the study. This way will be patients blinded.

Second examination will be provided after 6 months. Patients will be in the beginning introduced to doctor only by their unique number. Doctor will be blinded and he will not dispose with information about microinvasive procedure and will examine patient. Data which will be collected: (Visual analogue scale, pain radiating dermatome, global pain scale, changes in analgesics drugs consumption). All acquired information will be noted in to the special anonymous protocol. Also patients will anonymously fulfill Oswestry Low Back Disability Questionnaire. The third examination will be provided after 12 months same way. Patients will be in the beginning introduced to doctor only by their unique number. Doctor will be blinded and he will not dispose with information about microinvasive procedure and will examine patient. Data which will be collected: (Visual analogue scale, dermatome where pain is radiating, global pain scale, changes in analgesics drugs consumption). All acquired information will be noted in to the special anonymous protocol. Also patients will anonymously fulfill Oswestry Low Back Disability Questionnaire (ODI). If the patient will need to a see a doctor in the reason of deterioration of pain feeling and if the ODI will not increase more than 10% against patient's origin ODI value than one PRT is allowed in the spinal space responding to a pain radiating dermatome during first six months after patients inclusion to trial. Under the same conditions another PRT is allowed during next six months.

When ODI will increase more than 10% against patient's origin ODI value and more than 1 PRT during six month interval will be needed, than patient will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older
* Written informed consent
* Herniated disc, nerve compression, radicular syndromes (vertebrogenic algic syndrome)
* magnetic resonance examination evidence of intervertebral disc herniation
* Pain radiating to the lower limbs
* Disc lesion one level higher than dermatome with pain symptoms

Exclusion Criteria:

* Patients not capable of consenting
* pregnant women or women of child-bearing potential
* Previous spine operations
* Protrusion of more than one intervertebral disc
* Cauda equine syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Pain as assessed by the Visual analogue scale | 3 years
  All acquired information will be noted in to the special anonymous protocol

SECONDARY OUTCOMES:
Pain progress as assessed by global pain scale | 3 years
  All acquired information will be noted in to the special anonymous protocol
Changes in analgesics drugs consumption as assessed by equianalgesic dose ratios for opioids | 3 years
  All acquired information will be noted in to the special anonymous protocol
Pain localization as assessed by note of radiating dermatome as neurologic examination | 3 years
  All acquired information will be noted in to the special anonymous protocol
Number of extra PRT procedures | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Juraj Mláka, MD PhD, Study Chair — R-Clinic jmlaka@gmail.com
Locations (2):
- Czechia (2):
  - Algesiology ambulance, Prague, Czech Republic
  - Czech republic, Prague

REFERENCES:
- See also: website — http://www.europainclinics.com/